CLINICAL TRIAL: NCT00272454
Title: The Double-Blind, Randomized, Multi-Center, and Active Controlled Trial for Efficacy and Safety of Cilostazol in Acute Ischemic Stroke
Brief Title: Cilostazol in Acute Ischemic Stroke Treatment (CAIST)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Seoul National University Boramae Hospital (Other); Korea Otsuka International Asia Arab Co., Ltd. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOP-PLT-0501; NCT00272129 (obsolete NCT alias)
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Cerebral Infarction
Keywords: cilostazol; aspirin; cerebral infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — Cilostazol; Aspirin

INTERVENTIONS:
Drug: Cilostazol
Drug: Aspirin

SUMMARY:
The purpose of this study is to study efficacy and safety of cilostazol use in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and elderly disability in developed countries. However, treatment of acute stroke is limited except thrombolytic therapy in hyperacute stroke within several hours. Currently, aspirin is widely used in spite of its small benefit compared to bleeding complications.

Cilostazol will be compared to aspirin in acute stroke patients in terms of functional outcome at 3 months, efficacy to prevent stroke recurrence, and safety for bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive explanation on this study and give informed consent
* Patients aged 30 to 85 years
* Baseline NIHSS less than 15
* Onset of symptoms within 48 hours of the start of investigational product
* Full functional independence prior to the present stroke indicated by an mRS score of 0, 1, 2

Exclusion Criteria:

* Evidence from CT or MRI scan of an acute intracranial hemorrhage, a tumor, encephalitis or any diagnosis other than acute ischemic stroke likely to cause the present symptoms.
* Previous regular use of an antiplatelet agent or warfarin
* Patients with known cardiac disease likely to cause cardiogenic embolism or congestive heart failure
* Evidence from CT or MRI scan of midline shift when visiting hospital
* Uncontrolled hypertension (SBP>220 mmHg or DBP>120 mmHg)
* Hypotension (<90/60 mmHg)
* Patients with known bleeding diathesis or coagulation disorder
* Patients with liver disease (ALT>100 or AST>100), or renal disease (creatinine>2.0 mg/dl)
* Known severe anaemia (hemoglobin<8.0 mg/dl), or thrombocytopenia (platelet<100,000/mm3)
* Scheduled for endarterectomy within 3 months
* Severe co-morbidity likely to limit patient's life expectancy to less than 6 months
* Patients with alcohol or illegal drug abuse or dependency
* Pregnant or lactating patients. When administrating to females, it should be confirmed that the patients is in the menopause (by evaluation of investigators) or permanently infertile (hysterectomy or surgical operation like bilateral tubal ligation, bilateral oophorectomy, etc). If a patient is likely to be pregnant, the patient should not be pregnant before randomization. And, the patient should use reliable contraception between at least 3 weeks before randomization to 7 days after the final administration of study drug.
* Patients treated by thrombolytic agents like tPA after onset of stroke

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2006-01; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the frequency of mRS 0, 1, 2 at 90 days | at 90 days

SECONDARY OUTCOMES:
Frequency of mRS 0,1 at 90 days | at 90 days
Frequency of Barthel index 95-100 at 90 days
Frequency of mRS 0,1 & Barthel index 95-100 at 90 days
Frequency of NIHSS 0-1 at 90 days
Frequency of progression of neurological deficit at 7 days (increment of NIHSS 2 points or a point on the item of upper or lower extremity weakness)
Bleeding disorders (life-threatening bleeding; major bleeding; minor Bleeding)
Overall cardiovascular events (Ischemic heart disease requiring rehospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Seok Lee, M.D., PhD, Principal Investigator — Department of Neurology, Seoul National University Boramae Hospital, College of Medicine, Seoul National University
Locations (12):
- South Korea (12):
  - Hallym University Sacred Heart Hospital, Ahnyang, Kyunggi Province
  - Inje University Ilsan Paik Hospital, Koyang, Kyunggi Province
  - Seoul National University Bundang Hospital, Sungnam, Kyunggi Province
  - Eulji University Hospital, Daejeon
  - Inha University Hospital, Incheon
  - Dongguk University Hospital, Koyang, Kyunggi Province
  - Seoul National University Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Asan Medical Center, Seoul
  - Eulji University Hospital, Seoul
  - Seoul National University Boramae Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul

REFERENCES:
- [Derived] Lee YS, Bae HJ, Kang DW, Lee SH, Yu K, Park JM, Cho YJ, Hong KS, Kim DE, Kwon SU, Lee KB, Rha JH, Koo J, Han MG, Lee SJ, Lee JH, Jung SW, Lee BC, Kim JS. Cilostazol in Acute Ischemic Stroke Treatment (CAIST Trial): a randomized double-blind non-inferiority trial. Cerebrovasc Dis. 2011;32(1):65-71. doi: 10.1159/000327036. Epub 2011 May 25. PMID 21613787